CLINICAL TRIAL: NCT02203487
Title: A Double-blind (Within Dose Groups), Randomised, Placebo-controlled, Parallel-group Study to Investigate the Safety, Tolerability and Preliminary Pharmacokinetics of Increasing Repeated Oral Doses (Nine Days Treatment of 5 mg and 10 mg and Eighteen Days Treatment of 25 mg and 40 mg) of BIIF 1149 BS in Healthy Male Volunteers
Brief Title: Safety, Tolerability and Pharmacokinetics of Increasing Repeated Doses of BIIF 1149 BS in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1157.3
Record Dates: First submitted 2014-07-29; First posted 2014-07-30 (Estimated); Last update posted 2014-07-30 (Estimated); Status verified 2014-07

CONDITIONS: Healthy

ARMS (2):
- BIIF 1149 BS - single rising dose (Experimental)
  Interventions: Drug: BIIF 1149 BS - single rising dose
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIIF 1149 BS - single rising dose
  Arms: BIIF 1149 BS - single rising dose
Drug: Placebo
  Arms: Placebo

SUMMARY:
The objective of the present study was to obtain information about the safety and tolerability of BIIF 1149 BS after repeated dosing and to obtain preliminary pharmacokinetics data (steady state and accumulation factor)

ELIGIBILITY:
Inclusion Criteria:

* Participants should be healthy males
* Age range from 21 to 50 years
* Within +- 20% of their normal weight (Broca-Index)
* In accordance with Good Clinical Practice (GCP) and local legislation each volunteers are supposed to give their written informed consent prior to admission to the study
* Each subject will have his medical history taken and will receive a complete medical examination (incl. demographics, medical history, check of inclusion/exclusion criteria, physical examination, vital signs, 12-lead Electrocardiogram (ECG)
* Haematopoietic, hepatic and renal function test will be carried out in the laboratory
* The subjects will fast for 12 hours before collection of specimens for all laboratory evaluations. The above mentioned examinations will be performed within 14 days before the first administration of the test substance

Exclusion Criteria:

* Volunteers will be excluded from the study if the results of the medical examination or laboratory tests are judged by the clinical investigator to differ significantly from normal clinical values
* Volunteers with known gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Volunteers with diseases of the central nervous system (such as epilepsy) or with psychiatric disorders
* History of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of a drug with a long half-life (>= 24 hours) within ten half-lives of the respective drug before enrolment in the study
* Use of any other drugs which might influence the results of the trial during the week previous to the start of the study
* Participation in another study with an investigational drug within the last two months preceding this study
* Smoker (> 10 cigarettes or 3 cigars or 3 pipes/day)
* Inability to refrain from smoking on study days
* Alcohol abuse (> 40g/day)
* Drug abuse
* Blood donation (>= 100 ml) within the last 4 weeks
* Excessive physical activities (e.g. competitive sports) within the last week before the study

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 1999-11; Primary Completion 2000-06 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events | up to 55 days
Number of subjects with abnormal changes in laboratory parameters | up to 8 days after last blood sample
Number of subjects with clinically significant changes in vital signs (blood pressure, pulse rate) | up to 8 days after last blood sample

SECONDARY OUTCOMES:
Number of subjects with clinically significant changes in 12-lead Electrocardiogram (ECG) | up to 8 days after last blood sample
Cmax (Maximum concentration of the analyte in plasma) | up to 360 hours after last drug administration
Tmax (Time to maximum observed concentration of the analyte in plasma) | up to 360 hours after last drug administration
AUC (Area under the concentration-time curve of the analyte in plasma) | up to 360 hours after last drug administration
Ae (Urinary excretion of parent drug) | up to 120 hours after last drug administration
Cmin,ss (Minimum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ) | after 24 hours of drug administration on day 9
MRT (Mean residence time of the analyte in the body) | up to 360 hours after last drug administration
t½ (Terminal half-life of the analyte in plasma) | up to 360 hours after last drug administration
Percent peak-trough fluctuation | up to 360 hours after last drug administration
RA (AUC) Accumulation factor based on AUC-data | up to 360 hours after last drug administration
RA (Ae) Accumulation factor based on Ae-data | up to 120 hours after last drug administration
RA (Cmax) Accumulation factor based on Cmax -data | up to 360 hours after drug administration on day 9
Cav (Average plasma concentration in a steady state interval) | 24 hours after drug administration of day 9